## Breaking Down Care Process and Patient-level Barriers to Arteriovenous Access Creation Prior to Hemodialysis Initiation

Clinical Trials # NCT04032613 Principal Investigator: Jennifer E. Flythe Funded by: NIH/ NIDDK

> Statistical Analysis Plan Version Date: July 19th, 2019

Study participants will complete pre-program implementation and post-program implementation questionnaires to assess the effect of the program on their knowledge of dialysis vascular access and confidence navigating the dialysis vascular access creation process. We will use a paired sample student's t-test to compare participants' pre-program implementation and post-program implementation questionnaire scores. Analyses will be performed in SAS v9.4 and R v3.3.2 or later. Questionnaires are found in the study protocol.